CLINICAL TRIAL: NCT00181545
Title: Individualised Radiation Dose Determination on Basis of Normal Tissue Dose Constraints in Patients With Non-Small-Cell Lung Cancer: A Phase I Study
Brief Title: Safety Study of Individualised Radiation Dose Determination for Lung Cancer Patients.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04.1338L; MAASTRO 04-06
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Non-small cell lung carcinoma; radiotherapy; mean lung dose
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: escalation of dose (radiotherapy treatment)

SUMMARY:
Radiotherapy is treatment of choice for inoperable lung cancer. Research has shown that the local control rate is low and the radiation often causes pneumonitis and/or esophagitis.

To predict to lung damage the mean lung dose can be calculated. This allows us to give a higher total dose to the tumor and to improve the local control rate.

Study hypothesis: It will be safe to administer a radiation dose as high as possible to the tumor, taking into account the mean lung dose, calculated by the treatment planning system.

DETAILED DESCRIPTION:
Radiotherapy is treatment of choice for inoperable lung cancer. Research has shown that the survival rate as well as the local control rate is low. If chemotherapy treatment is added it leads to a slightly better outcome. The radiotherapy treatment often causes pneumonitis and/or esophagitis. So damage to the normal tissue restricts the radiation dose that can be administered.

However, several studies have shown that higher doses lead to better local control. Furthermore it is evident that the radiotherapy treatment should be given in a short time, preferably the treatment time should not exceed 32 days.

To avoid a higher toxicity the normal tissue has to be spared, but to increase the local control rate the tumor dose must be as high as possible. This dilemma can only be solved by using very sophisticated treatment planning techniques in combination with a biologically superior treatment schedule. This schedule consists of delivering radiation dose twice a day instead of once, thus keeping the overall treatment time as low as possible.

For the whole patient population, the mean lung dose can to a great extend predict the probability for developing radiation pneumonitis and the post-radiotherapy lung function. A logical next step is to determine the dose of radiotherapy on an individualised calculation of the maximum tolerated dose, being defined as the mean lung dose and the spinal cord dose.

The objective of this trial is to investigate whether individualised radiation dose calculation based on a mean lung dose and the constraints of the spinal cord, in combination with an overall treatment time of less than 32 days, and only irradiating the primary tumor and the PET scan positive mediastinal areas is safe.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-small cell lung cancer
* UICC stage I-III
* WHO performance status 0-2
* Less than 10 % weight loss the last 6 months
* In case of previous chemotherapy, radiotherapy can start after a minimum of 21 days after the last chemotherapy course
* Reasonable lung function: FEV1 ³ 60 % of the predicted value
* No recent ( < 3 months) severe cardiac disease (arrhythmia, congestive heart failure, infarction)
* No active peptic oesophagitis
* Life expectancy more than 6 months
* Measurable cancer
* Willing and able to comply with the study prescriptions
* 18 years or older
* Not pregnant and willing to take adequate contraceptive measures during the study
* Have given written informed consent before patient registration
* No previous radiotherapy to the chest

Exclusion Criteria:

* Not non-small cell histology, e.g. mesothelioma, lymphoma
* Mixed pathology, e.g. non-small cell plus small cell cancer
* Malignant pleural or pericardial effusion
* Concurrent chemotherapy with radiation
* History of prior chest radiotherapy
* Recent ( < 3 months) myocardial infarction
* Uncontrolled infectious disease
* Distant metastases (stage IV)
* Patients with active peptic oesophagitis in the last year.
* Less than 18 years old
* Pregnant or not willing to take adequate contraceptive measures during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
incidence of steroid dependent (grade 2 or more) radiation pneumonitis 6 months after the last radiotherapy dose.

SECONDARY OUTCOMES:
incidence of radiation pneumonitis according to the location of the primary tumour
acute esophagitis
FEV1 6 months after radiotherapy
DLCO 6 months after radiotherapy
late esophagitis, 6 months after radiotherapy
tumor response, 70 days post chest radiotherapy
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, PHD, Principal Investigator — Maastricht Radiation Oncology (MAASTRO clinic)
Locations (1):
- Maastircht Radiation Oncology, Heerlen, Limburg, Netherlands